CLINICAL TRIAL: NCT03832036
Title: The Diagnostic and Prognostic Value of Two Quantitative Clinical Tests in Patients
Brief Title: The Diagnostic and Prognostic Value of Two Quantitative Clinical Tests in Patients With Lumbar Disc Herniation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Spine Centre of Southern Denmark (Other)
Collaborators: Frederiksberg University Hospital (Other); Center for Rheumatology and Spine Diseases, Frederiksberg Hospital, Denmark (Unknown); Odense University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 201170138
Record Dates: First submitted 2018-10-26; First posted 2019-02-06 (Actual); Last update posted 2025-07-08 (Actual); Status verified 2025-07

CONDITIONS: Pain; Lumbar Disc Herniation; Back Pain; Spinal Diseases; Surgery
Keywords: Electromyography; Paraspinal Mapping; Quantitative clinical tests; Conditioned pain modulation; Temporal pain summation; Pain threshold; Pain tolerance
MeSH Terms: conditions — Pain; Intervertebral Disc Displacement; Back Pain; Spinal Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients with lumbar disc herniation (Experimental)
  Interventions: Diagnostic Test: Paraspinal Mapping and Quantitative Sensory Pain Test

INTERVENTIONS:
Diagnostic Test: Paraspinal Mapping and Quantitative Sensory Pain Test — Participants will be tested at baseline.

SUMMARY:
This study will investigate whether two clinical tests can be used to diagnose and predict the outcome in patients with lumbar disc herniation undergoing surgery and non-surgery treatment.

The two quantitative clinical tests include: electromyographic measurements using Paraspinal Mapping and pain responses using Quantitative Sensory Pain Testing.

DETAILED DESCRIPTION:
150 patients will be included for the prospective cohort study. Patients will be recruited from the Region of Southern Denmark and Capital Region. Participants will undergo MRI scanning of the lumbar spine, fillout a questionnaire and undergo assessment with the two clinical tests. An 8-week follow-up will be made with patients completing a questionnaire. The two quantitative clinical tests include: electromyographic measurements using Paraspinal Mapping and pain responses using Quantitative Sensory Pain Testing.

ELIGIBILITY:
Inclusion Criteria:

* Clinical and radiologically diagnosed lumbar disc herniation.
* Low back pain with pain below the knee or anterior thigh pain in one or both legs.
* Dermatomal leg pain.
* Average pain intensity of 3 or more on a Numerical Rating Scale (0-10 NRS).

Exclusion Criteria:

* History of previous lumbar spine surgery.
* Surgery in general in the past 4 months.
* Current use of anticoagulants.
* Diagnoses which could confound with the diagnosis e.g. lumbar spinal stenosis, local muscle trauma, cancer metastases, fibromyalgia, neuropathy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 102 (Actual)
Dates: Start 2018-10-01 (Actual); Primary Completion 2021-01-01 (Actual); Study Completion 2021-01-01 (Actual)

PRIMARY OUTCOMES:
The diagnostic value of Paraspinal Mapping and Quantitative Sensory Pain Testing | 8 week follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Johanne B Filtenborg, M.Sc., Principal Investigator — Spine Centre Southern Denmark; Berit Schiøttz-Christensen, MD, Study Director — Spine Centre Southern Denmark; Søren O'Neill, DC, Study Chair — Spine Centre Southern Denmark; Kirstine Amris, MD, Study Chair — The Parker Institute, Frederiksberg Hospital; Gilles Fournier, MD, DC, Study Chair — Center for Rheumatology and Spine Diseases, Frederiksberg Hospital; Andrew J Haig, MD, Study Chair — University of Michigan
Locations (1):
- Center for Rheumatology and Spine Diseases, Frederiksberg Hospital., Frederiksberg, Denmark

IPD SHARING:
Plan to Share IPD: Undecided

DOCUMENTS (1):
  • Statistical Analysis Plan (2023-06-27): https://cdn.clinicaltrials.gov/large-docs/36/NCT03832036/SAP_001.pdf